CLINICAL TRIAL: NCT00646997
Title: Impact Of Velocity Vector Imaging, Tissue Doppler Imaging, Conventional Echocardiography And P Wave Dispertion In Evaluating Post-Operative Atrial Fibrillation After Coronary Bypass Graft Surgery
Brief Title: Impact of Left Atrial Function on Postoperative Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Prof.Dr.Saide Aytekin, T.C. Istanbul Bilim University, Florence Nightingale Hospital
Other Study IDs: YT1977/2
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, left atrium, velocity vector imaging
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with postoperative atrial fibrillation
- 2: Patients without postoperative atrial fibrillation.

SUMMARY:
We aimed to demonstrate the impact of left atrial functions which were evaluated by three different echocardiographic modalities , on postoperative atrial fibrillation.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation after coronary artery bypass greft operation (CABG) is major complication with a prevalence of 10-50%. Although the men mechanism is not known, in recent studies, age and left atrial function have been demonstrated as the most responsible factors. Velocity vector imaging (VVI) is a new modality which may give accurate and detailed information on both left atrial segmental and global function. In this study, our aim was to assess preoperative left atrial function by using three different echocardiographic modalities, VVI, tissue Doppler imaging and conventional echocardiography and evaluate the relation between the left atrial functions and the development of post-operative atrial fibrillation after CABG.

ELIGIBILITY:
Inclusion Criteria:

* 1Coronary artery disease evidenced by coronary angiography
* 2Patients with a decision of undergoing elective coronary artery bypass greft operation
* 3Sinus rhythm in electrocardiography

Exclusion Criteria:

* 1Rheumatic valve disease
* 2Having prosthetic valve
* 3CABG accompanied by other cardiac interventions (such as valvular surgery, ASD closure...etc)
* 4Left ventricular l ejection fraction <40%
* 5Mild to moderate mitral stenosis or regurgitation
* 6Having atrial fibrillation or a history of atrial fibrillation attach during the last two weeks.
* 7Congenital heart disease
* 8Chronic liver disease
* 9Chronic renal disease
* 10Malignancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Velocity vector imaging derived left atrial segmenter function, Tissue doppler derved left atrial segmenter function, conventional analysis of atrial function by 2D and pulsed wave echocardiography. | April 2008

CONTACTS AND LOCATIONS:
Overall Officials: Saide Aytekin, Professor, Study Director — T.C. Istanbul Bilim University, Florence Nightingale Hospital, Division of Cardiology
Locations (1):
- TC.Istanbul Bilim University, Florence Nightingale Hospital, Division of Cardiology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] 1-Leung JM, Bellows WH, Schiller NB. Impairment of left atrial function predicts post-operative atrial fibrillation after coronary artery bypass graft surgery. European H J. 2004,25,1836-1844 2-Nakai T , Lee R, Schiller N, et al. The relative importance of left atrial function versus dimension in predicting atrial fibrilation after coronary bypass graft surgery. Am H Journal. 2002; 143:181-6